CLINICAL TRIAL: NCT00955721
Title: A Phase I/II Study of Combination of Gemcitabine, Oxaliplatin and Sorafenib (GEMOX-Sorafenib) in Patients With Advanced Biliary Tract Cancer
Brief Title: A Study of Combination of Gemcitabine, Oxaliplatin (GEMOX)-Sorafenib in Patients With Advanced Biliary Tract Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of Funding
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Peter Hosein, Assistant Professor of Clinical, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20090256; SCCC-2009003 (Other: UM/Sylvester Comprehensive Cancer Center)
Record Dates: First submitted 2009-08-06; First posted 2009-08-10 (Estimated); Results first posted 2015-02-13 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Cholangiocarcinoma; Biliary Tract Cancer; Gallbladder Cancer
Keywords: Cholangiocarcinoma; Biliary Tract Cancer; Gallbladder Cancer
MeSH Terms: conditions — Cholangiocarcinoma; Biliary Tract Neoplasms; Gallbladder Neoplasms | interventions — Gemcitabine; Oxaliplatin; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase 1: GEMOX + Sorafenib (Experimental): Gemcitabine and Oxaliplatin (GEMOX) and Sorafenib.
  * Gemcitabine: 1000 or 750 mg/m2, IV, Day 1 of each 14 day cycle, until progression or unacceptable toxicity develops.
  * Oxaliplatin: 100 or 75 mg/m2, IV, Day 2 of each 14 day cycle, until progression or unacceptable toxicity develops.
  * Sorafenib: 200 mg, Orally, twice daily for each 14-day cycle, until progression or unacceptable toxicity develops.
  Interventions: Drug: Gemcitabine; Drug: Oxaliplatin; Drug: Sorafenib
- Phase 2 - RPTD GEMOX + Sorafenib (Experimental): Recommended Phase Two Dose (RPTD) of Gemcitabine and Oxaliplatin (GEMOX) and Sorafenib:
  * Gemcitabine: Recommended Phase II Dose determined from Phase I, Day 1 of each 14 day cycle, until progression or unacceptable toxicity develops.
  * Oxaliplatin: Recommended Phase II Dose determined from Phase I, Day 2 of each 14 day cycle, until progression or unacceptable toxicity develops.
  * Sorafenib: Recommended Phase II Dose determined from Phase I, Orally, twice daily for each 14-day cycle, until progression or unacceptable toxicity develops.
  Interventions: Drug: Gemcitabine; Drug: Oxaliplatin; Drug: Sorafenib

INTERVENTIONS:
Drug: Gemcitabine — Intravenously (IV) on Day 1 of each 14 day cycle, until progression or unacceptable toxicity develops.
  Other Names: Gemzar
Drug: Oxaliplatin — Intravenously (IV) on Day 2 of each 14 day cycle, until progression or unacceptable toxicity develops.
  Other Names: Eloxatin
Drug: Sorafenib — Orally, twice daily for each 14-day cycle, until progression or unacceptable toxicity develops.
  Other Names: BAY 43-9006

SUMMARY:
The purpose of this study is to build on the efficacy of the GEMOX regimen by adding Sorafenib in the treatment of Biliary Tract Cancer. Since there is no data on the combination of these three agents, the investigators plan to evaluate the safety in a run-in phase I portion in order to define the recommended phase II dose (RPTD). The phase II trial will enroll 40 patients at the RPTD level within 2 years in order to provide a preliminary estimate of progression-free survival (primary endpoint of the trial) in the target population.

DETAILED DESCRIPTION:
The purpose of this study is to build on the efficacy of the GEMOX regimen by adding Sorafenib in the treatment of Biliary Tract Cancer. Since there are no data on the combination of these three agents, the investigators plan to evaluate the safety in a run-in phase I portion in order to define the recommended phase II dose (RPTD). The phase II trial will enroll 40 patients at the RPTD level within 2 years in order to provide a preliminary estimate of progression-free survival (primary endpoint of the trial) in the target population.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Histologically or cytologically confirmed biliary tract or gallbladder carcinoma
* Any stage of disease is allowed but the patients must not be candidates for curative resection
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1 in Ph I
* ECOG performance status 0-2 in Ph II. Patients with ECOG PS of 2 will only be enrolled if they will comprise at most 25% of the total accruals. This will be monitored in real time to ensure that at any point during accrual, PS 2 patients will comprise <= 25% of the total accruals
* Patients must have normal organ and marrow function as defined below within 14 days of study entry:

  * Absolute neutrophil count >= 1,500 cells/mm3
  * Platelet count >= 60,000/mm3
  * Creatinine < 1.5 upper limit of normal (ULN).
  * Aspartate transaminase (AST) and Alanine transaminase (ALT) <= 2.5 x ULN.
  * Bilirubin <= 3.0 mg/dl
  * International normalized ratio (INR) < 1.5 or a prothrombin time (PT)/partial thromboplastin time (PTT) within normal limits. Patients receiving anti-coagulation treatment with an agent such as warfarin will not be candidates for the trial. Patients on anticoagulation with low molecular weight or heparinoids are protocol candidates.
* Any number of previous lines of chemotherapy is allowed for the phase I portion
* During the phase II trial, no prior chemotherapy for inoperable or metastatic disease is allowed except 5-FU or Capecitabine as radiosensitizers. Prior adjuvant chemotherapy is allowed.
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment
* Women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation. Men should use adequate birth control for at least three months after the last administration of sorafenib.
* Ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained prior to any study specific procedures.
* Life expectancy of greater than 12 weeks

Exclusion Criteria:

* Investigational agents within 28 days prior to Day 1 of study
* Chemotherapy within 4 weeks prior to Day 1 of study
* Nitrosoureas, mitomycin-C within 6 weeks prior to Day 1 of study.
* Prior treatment with sorafenib, gemcitabine or oxaliplatin
* Prior history of peripheral neuropathy > Grade 1 (e.g., diabetic neuropathy)
* Pregnant or breast-feeding female
* Patients with a history of allergic reactions or sensitivity attributed to compounds of similar chemical or biologic composition to sorafenib, oxaliplatin or gemcitabine
* Patients with GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis)
* Cardiac disease: Congestive heart failure > class II New York Heart Association (NYHA). Patients must not have unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
* Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management.
* Known brain metastasis. Patients with neurological symptoms must undergo a CT scan/MRI of the brain to exclude brain metastasis.
* Known human immunodeficiency virus (HIV) infection and Hepatitis B and Hepatitis C.
* Active clinically serious infection > CTCAE Grade 2.
* Arterial thrombotic/embolic events like myocardial infarct and cerebrovascular accident including transient ischemic attacks within the past 6 months.
* Pulmonary hemorrhage/bleeding event > CTCAE Grade 2 within 4 weeks of first dose of study drug.
* Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug.
* Serious non-healing wound, ulcer, or bone fracture.
* Evidence or history of bleeding diathesis or coagulopathy
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of first study drug.
* Use of St. John's Wort or rifampin (rifampicin).
* Any medical condition, which in the opinion of the investigator places the patient at an unacceptably high risk for toxicities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hosein, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: GEMOX + Sorafenib: Gemcitabine and Oxaliplatin (GEMOX) and Sorafenib:
  * Gemcitabine: 1000 or 750 mg/m2, IV, Day 1 of each 14 day cycle, until progression or unacceptable toxicity develops.
  * Oxaliplatin: 100 or 75 mg/m2, IV, Day 2 of each 14 day cycle, until progression or unacceptable toxicity develops.
  * Sorafenib: 200 mg, Orally, twice daily for each 14-day cycle, until progression or unacceptable toxicity develops.
- Phase 2: RPTD GEMOX + Sorafenib: Recommended Phase Two Dose (RPTD) of Gemcitabine and Oxaliplatin (GEMOX) and Sorafenib:
  * Gemcitabine: Recommended Phase II Dose determined from Phase I, Day 1 of each 14 day cycle, until progression or unacceptable toxicity develops.
  * Oxaliplatin: Recommended Phase II Dose determined from Phase I, Day 2 of each 14 day cycle, until progression or unacceptable toxicity develops.
  * Sorafenib: Recommended Phase II Dose determined from Phase I, Orally, twice daily for each 14-day cycle, until progression or unacceptable toxicity develops.
Period: Overall Study
Arm/Group | Phase 1: GEMOX + Sorafenib | Phase 2: RPTD GEMOX + Sorafenib
Started | 9 | 0
Completed | 6 | 0
Not Completed | 3 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: GEMOX + Sorafenib | Phase 2: RPTD GEMOX + Sorafenib | Total
Number analyzed (Participants) | 9 | 0 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 2 |  | 2
  >=65 years | 7 |  | 7
Age, Continuous [Mean (Full Range); unit: years] | 67.4 [59 to 74] |  | 67.4 [59 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 |  | 3
  Male | 6 |  | 6
Region of Enrollment [Number; unit: participants]
  United States | 9 |  | 9

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Recommended Phase II Dose (RPTD) of the Combination of Sorafenib and GEMOX in Patients With Advanced Biliary Tract Cancer (BTC).
Description: Establish the recommended phase II dose (RPTD) of the combination of sorafenib and GEMOX in patients with advanced biliary tract cancer (BTC).
Time Frame: First two 14-day Phase I cycles
Population: A total of 9 participants were enrolled in Phase 1 of which 6 were evaluable and analyzed for this outcome measure. A recommended phase two dose (RPTD) of the combination of Sorafenib and GEMOX therapy could not be determined because dose escalation was still in progress when the study was terminated.
Measure: Number; unit: mg
Groups:
- Phase 1: GEMOX + Sorafenib: Gemcitabine and Oxaliplatin (GEMOX) and Sorafenib.
  * Gemcitabine: 1000 or 750 mg/m2, IV, Day 1 of each 14 day cycle, until progression or unacceptable toxicity develops.
  * Oxaliplatin: 100 or 75 mg/m2, IV, Day 2 of each 14 day cycle, until progression or unacceptable toxicity develops.
  * Sorafenib: 200 mg, Orally, twice daily for each 14-day cycle, until progression or unacceptable toxicity develops.
  Gemcitabine: Intravenously (IV) on Day 1 of each 14 day cycle, until progression or unacceptable toxicity develops.
  Oxaliplatin: Intravenously (IV) on Day 2 of each 14 day cycle, until progression or unacceptable toxicity develops.
  Sorafenib: Orally, twice daily for each 14-day cycle, until progression or unacceptable toxicity develops.
Arm/Group | Phase 1: GEMOX + Sorafenib
Number analyzed (Participants) | 6
mg
  Gemcitabine | NA — A recommended phase two dose (RPTD) of the combination of Sorafenib and GEMOX therapy could not be determined because dose escalation was still in progress when the study was terminated.
  Oxaliplatin | NA — A recommended phase two dose (RPTD) of the combination of Sorafenib and GEMOX therapy could not be determined because dose escalation was still in progress when the study was terminated.
  Sorafenib | NA — A recommended phase two dose (RPTD) of the combination of Sorafenib and GEMOX therapy could not be determined because dose escalation was still in progress when the study was terminated.

2. Primary Outcome: Phase II: Obtain an Estimate of the 9-month Progression-free Survival Rate in Patients With Advanced BTC Receiving the RPTD of the Combination Sorafenib and GEMOX.
Description: Rate of study participants achieving progression-free survival at 9 months post-initiation of study therapy at RPTD. Progression-Free Survival (PFS) is defined as the time elapsed from the start of treatment to the date of documented progression or death, whichever comes first. For surviving patients without progression who begin alternative treatment, PFS will be censored at the last date of documented progression-free status prior to starting alternative treatment. Similarly, losses to follow up will be censored at the last date of documented progression-free status.
Time Frame: 9 Months
Population: This was an outcome measure for the Phase 2 arm. Data were not collected due to the study's termination prior to the determination of the RPTD and the opening of Phase 2.
Arm/Group | Phase 2: RPTD GEMOX + Sorafenib
Number analyzed (Participants) | 0

3. Secondary Outcome: Phase II: Estimate Overall Response Rate and Clinical Benefit Rate.
Description: Overall response rate [CR + PR]. Clinical Benefit Rate [Complete Response (CR) + Partial Response (PR) + Stable Disease (SD)] per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0).
Time Frame: About 9 Months
Population: This was an outcome measure for the Phase 2 arm. Data were not collected due to the study's termination prior to the opening of Phase 2.
Arm/Group | Phase 2: RPTD GEMOX + Sorafenib
Number analyzed (Participants) | 0

4. Secondary Outcome: Phase II: Estimate Overall Survival
Description: Overall survival is defined as the time elapsed from the start of treatment until death. For surviving patients, follow-up will be censored at the date of last contact.
Time Frame: Start of treatment until death or date of last contact
Population: as for outcome 3
Groups:
- Phase 2 - RPTD GEMOX + Sorafenib: Recommended Phase Two Dose (RPTD) of Gemcitabine and Oxaliplatin (GEMOX) and Sorafenib:
  * Gemcitabine: Recommended Phase II Dose determined from Phase I, Day 1 of each 14 day cycle, until progression or unacceptable toxicity develops.
  * Oxaliplatin: Recommended Phase II Dose determined from Phase I, Day 2 of each 14 day cycle, until progression or unacceptable toxicity develops.
  * Sorafenib: Recommended Phase II Dose determined from Phase I, Orally, twice daily for each 14-day cycle, until progression or unacceptable toxicity develops.
  Gemcitabine: Intravenously (IV) on Day 1 of each 14 day cycle, until progression or unacceptable toxicity develops.
  Oxaliplatin: Intravenously (IV) on Day 2 of each 14 day cycle, until progression or unacceptable toxicity develops.
  Sorafenib: Orally, twice daily for each 14-day cycle, until progression or unacceptable toxicity develops.
Arm/Group | Phase 2 - RPTD GEMOX + Sorafenib
Number analyzed (Participants) | 0

5. Secondary Outcome: Phase II: Further Evaluate the Safety of the Proposed Combination
Description: Rate of study participants experiencing toxicity after receiving study therapy at the recommended Phase 2 Dose (RPTD).
Time Frame: About 9 Months
Population: as for outcome 3
Arm/Group | Phase 2 - RPTD GEMOX + Sorafenib
Number analyzed (Participants) | 0

6. Secondary Outcome: Phase II: Explore Biomarkers of Response to the Combination
Description: A study of the correlation between biomarker levels and response to RPTD study therapy. Blood samples for biomarker analysis are collected at baseline and on day 1 of Cycles 2 onward
Time Frame: Baseline, Day 1 of Cycle 2 and subsequent cycles, about 9 Months
Population: as for outcome 3
Arm/Group | Phase 2 - RPTD GEMOX + Sorafenib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Phase 1: GEMOX + Sorafenib | Phase 2: RPTD GEMOX + Sorafenib
All-Cause Mortality (participants affected / at risk) | 4/9 | 0/0
Serious Adverse Events (participants affected / at risk) | 3/9 | 0/0
Other Adverse Events (participants affected / at risk) | 8/9 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: GEMOX + Sorafenib (N=9) | Phase 2: RPTD GEMOX + Sorafenib (N=0)
Peritoneal Infection (Infections and infestations) | 1 (1) | 0 (0)
Dehydration (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (2) | 0 (0)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: GEMOX + Sorafenib (N=9) | Phase 2: RPTD GEMOX + Sorafenib (N=0)
Vomiting (Gastrointestinal disorders) | 4 (6) | 0 (0)
Vaginal Hemorrhage (Vascular disorders) | 1 (2) | 0 (0)
Urine Discoloration (Renal and urinary disorders) | 1 (1) | 0 (0)
Toothache (General disorders) | 1 (2) | 0 (0)
Taste Alteration (Gastrointestinal disorders) | 2 (2) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Rectal hemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (6) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 5 (13) | 0 (0)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 5 (17) | 0 (0)
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 6 (14) | 0 (0)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 7 (18) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Abdominal Distention (Gastrointestinal disorders) | 1 (2) | 0 (0)
Allergic Reaction (Immune system disorders) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Anorexia (Gastrointestinal disorders) | 6 (13) | 0 (0)
Anxiety (Nervous system disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Back Pain (General disorders) | 4 (6) | 0 (0)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (4) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Depression (Nervous system disorders) | 1 (1) | 0 (0)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Death - Disease Progression (General disorders) | 1 (1) | 0 (0)
Ear, nose and throat examination abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Edema limbs (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Fatigue (General disorders) | 7 (14) | 0 (0)
Fever (General disorders) | 2 (4) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
GI - Other (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Headache (General disorders) | 1 (1) | 0 (0)
Hearing (monitoring program) (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 8 (24) | 0 (0)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (11) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (5) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Hypertension (Cardiac disorders) | 3 (5) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (19) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (8) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (5) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (10) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Joint Pain (General disorders) | 2 (2) | 0 (0)
Leukocytes (Blood and lymphatic system disorders) | 6 (21) | 0 (0)
Liver dysfunction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 5 (11) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (9) | 0 (0)
Neutrophils (Blood and lymphatic system disorders) | 2 (8) | 0 (0)
Pain (General disorders) | 1 (2) | 0 (0)
Pain - Other (General disorders) | 3 (4) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (14) | 0 (0)
Pharyngolaryngeal pain (General disorders) | 2 (3) | 0 (0)
Platelets (Blood and lymphatic system disorders) | 6 (16) | 0 (0)

LIMITATIONS AND CAVEATS:
Study terminated due to lack of funding prior to the opening of the Phase 2 arm. Minimum required enrollment of 18 evaluable participants for Phase 1 not met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes